CLINICAL TRIAL: NCT02291991
Title: A Randomized, Double-blind Placebo Controlled, Single-dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of GX-E2 After Single Intravenous Administration in Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of GX-E2 in Healthy Subjects
Acronym: GX-E2-P1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GX-E2-P1
Record Dates: First submitted 2014-10-30; First posted 2014-11-17 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Immunogenecity
MeSH Terms: interventions — GC1113

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Drug : GX-E2 - Intravenously injection once day at dose 8 ug/kg Drug : Placebo
  (1 subject : GX-E2, 1 subject : Placebo)
  Subjects in group A will be injected drug, So we observe safety. After three days, Subject in group B will be injected drug.
  Interventions: Drug: GX-E2
- Group B (Experimental): Drug : GX-E2 - Intravenously injection once day at dose 8 ug/kg Drug : Placebo (7 subjects : GX-E2, 1 subject : Placebo)
  Interventions: Drug: GX-E2

INTERVENTIONS:
Drug: GX-E2 — Investigational drug(GX-E2 or Placebo) will be administered to healthy volunteers by the intravenous route.
  Other Names: GC1113
  Arms: Group A
Drug: GX-E2 — Investigational drug(GX-E2 or Placebo) will be administered to healthy volunteers by the intravenous route.
  Other Names: GC1113
  Arms: Group B

SUMMARY:
This is a randomized, placebo controlled, single dose study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of GX-E2 in healthy male subjects.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of GX-E2 when given as single dose (GX-E2 8 ug/kg) to healthy male subjects. Additionally, Immunogenecity will be evaluated to investigate antibody production.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male subjects 20 to 55 years old
* Adequate body weigth and BMI(19 ≤ BMI ≤ 27, 60.0kg ≤ body weigth ≤ 90.0kg)
* The subject doesn't have a clinically significant abnormal laboratory value and/or clinically significant unstable medical or disease history.
* Are eligible for the study hemoglobin data(12.0g/dL ≤ Hb ≤ 16.5g/dL) (Data is checked per 2 weeks within 28 days)
* Adequate transferrin saturation, serum ferritin within 28 days
* Adequate folate within 28 days
* Adequate vitamin B12 within 28 days
* Adequate WBC count (≥ 3.0 X 1000 µL)
* Adequate PLT count(≥ 140 X 1000 µL)
* nonsmoker or smoker smoked under 10 cigarettes a day

Exclusion Criteria:

* The subject has a clinically significant abnormal allergy including medical allergy.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease
* Subject with a previous experience in i.v. administration of EPO, darbepoetin, other EPO supplying proteins, immunoglobulin and iron drugs
* Subject with a hypersensitivity against EPO, darbepoetin and supplementary iron drugs
* Subject with a condition of hemoglobinopathy (e.g. sickle-cell disease and thalassemia)
* Subject showing following systolic and diastolic parameters at sitting position after 3 minutes of resting: lower than 90 mmHg or higher than 140mmHg of systolic blood pressure and lower than 50 mmHg or higher than 90mmHg of diastolic blood pressure
* Subject with chronic and uncontrollable symptoms of inflammatory disease (e.g. rheumatoid arthritis and systemic lupous erythematousus)
* Subject with the exceeding level of C-reactive protein more than 4 mg/dL before 2 weeks of IP administration
* History of drug prior to screening or urine drug testing is positive (cocaine, amphetamines, barbiturates, opiates, benzodiazepine, cannabinoids)
* Subject who has administered with a prescribed drug and oriental or herbal medicine in 2 weeks before IP administration, and who has administered with a general pharmaceutical and vitamin in 1 week before IP administration
* Subject who has enrolled in other clinical trials of IP or approved drug within 8 weeks before IP administration
* Subject with a history of fever at body temperature more than 38°C in a week before IP administration
* History of epileptic convulsion within 6 months
* Subject who is positive in HIV, HBsAg, HCV antibody test
* Subject with a regular alcohol consumption more than 21 unit, and who is unable to quit drinking during the period of clinical trial
* Subject who donated or lost more than 400mL of blood within 8 weeks prior to first dose
* Subject who is treated with investigational products.
* Subject with a longer length of spleen more than 16cm via upper abdominal ultrasound during the screening
* Subject who is considered as inappropriate for participation by Investigator based on various lab results
* Subject who plans to be pregnant or at least is unable to apply authorized contraceptive methods (e.g. sterilization operation, the use of contraceptive devices)

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics as measured by Cmax | Day1 - 29
  Measures "Cmax, AUC(0-tlast), AUCing, Tmax, t1/2 and CL/F after single dose of 8ug/kg GX-E2"
pharmacokinetics as measured by Cmax AUC(0-tlast) | Day1 - 29
  Measures "Cmax, AUC(0-tlast), AUCing, Tmax, t1/2 and CL/F after single dose of 8ug/kg GX-E2"
pharmacokinetics as measured by AUCing | Day1 - 29
  Measures "Cmax, AUC(0-tlast), AUCing, Tmax, t1/2 and CL/F after single dose of 8ug/kg GX-E2"
pharmacokinetics as measured by Tmax | Day1 - 29
  Measures "Cmax, AUC(0-tlast), AUCing, Tmax, t1/2 and CL/F after single dose of 8ug/kg GX-E2"
pharmacokinetics as measured by t1/2 | Day1 - 29
  Measures "Cmax, AUC(0-tlast), AUCing, Tmax, t1/2 and CL/F after single dose of 8ug/kg GX-E2"
pharmacokinetics as measured by CL/F | Day1 - 29
  Measures "Cmax, AUC(0-tlast), AUCing, Tmax, t1/2 and CL/F after single dose of 8ug/kg GX-E2"

SECONDARY OUTCOMES:
pharmacodynamics as measured by Hemoglobin | Day1 - 29
  Hemoglobin, Reticulocyte count, Reticulocyte hemoglobin contents
pharmacodynamics as measured by Reticulocyte count | Day1 - 29
pharmacodynamics as measured by Reticulocyte hemoglobin contents | Day1 - 29
Safety and Tolerability of GX-E2 as checked immunogenecity | Day1 - 29

CONTACTS AND LOCATIONS:
Overall Officials: KyungSang Yu, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea